CLINICAL TRIAL: NCT01067482
Title: The Performances of Spectral Domain Optical Coherence Tomography for Distinguishing Between Normal Eyes, Glaucoma Suspect and Glaucomatous Eyes
Brief Title: The Performances of Spectral Domain Optical Coherence Tomography (OCT) for Distinguishing Glaucomatous Eyes
Acronym: cirrusOCT
Status: Completed | Type: Observational
Sponsor: Prince of Songkla University (Other)
Responsible Party: Weerawat Kiddee, Glaucoma unit , Department of Ophthalmology Faculty of Medicine Prince of Songkla University Hat-yai,, Songkhla, Thailand., Thailand
Other Study IDs: EC 52-336-02-1-2
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2010-03-23 (Estimated); Status verified 2009-10

CONDITIONS: Glaucoma Patient; Glaucoma Suspect Patient; Normal Population; RNFL Thickness by Location; Macular Thickness by Location
Keywords: OCT; spectral domain cirrus; glaucoma; glaucoma suspect; normal population
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Glaucoma patients
- Glaucoma suspect group
- Normal population

SUMMARY:
The purpose of this study is to evaluate performances of each parameters of spectral domain (Cirrus) optical coherence tomography for distinguishing between normal eyes, glaucoma suspect and glaucomatous eyes

DETAILED DESCRIPTION:
Aim to determine which parameter of cirrus OCT is best sensitivity and specificity for glaucoma detection

ELIGIBILITY:
Inclusion Criteria:

* BCVA at least 20/60
* refractive error +/- 5 D Or astig +/- 3 D
* enrolled in 3 population group (glaucoma, glaucoma suspect or normal)

Exclusion Criteria:

* VA less than 20/60
* marked RF error
* previous ocular trauma or surgery
* unreliable visual field
* poor signal cirrus OCT (less than 7)
* other causes of optic nerve or macular disease other than glaucoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: glaucoma patient from glaucoma clinic that is POAG Glaucoma suspect cases normal population case
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Weerawat Kiddee, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- Glaucoma unit , Department of Ophthalmology Faculty of Medicine Prince of Songkla University, Hat Yai, Songkhla, Thailand., Thailand